CLINICAL TRIAL: NCT00457327
Title: Pilot Study for Evaluation of the Need for Protective Ileostomy After Low Anterior Resection Due to Rectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: RCT with same hypothesis ended and showed a superiority for protective ileostomy after lower anterior rectum resection.
Sponsor: Heidelberg University (Other)
Responsible Party: University of Heidelberg, Department of General, Visceral and Transplantation Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 433/2005
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Rectal Cancer
Keywords: protective ileostomy; rectal cancer; low anterior resection
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: protective ileostomy

SUMMARY:
The purpose of this study is to determine whether protective ileostomy is required after low anterior resection due to rectal cancer

DETAILED DESCRIPTION:
Since introduction of total mesorectal excision prognosis and quality of life of patients with rectal cancer of the middle or lower third of the rectum could be improved significantly. There is no valid data about the need of protective ileostomy in these patients. About 10% of the patients develop insufficiency of the anastomosis and might benefit from ileostomy whereas about 90% would not have required protective ileostomy retrospectively. Aim of the study is to show that protective ileostomy is not required if several criteria are fulfilled and early measures in case of clinical impairment are defined. Therefore eligibility criteria include safely performed stapler anastomosis with complete rings and control of impermeability by air insufflation. In the event of clinical impairment in the postoperative course CT scan with KM filling of the rectum to exclude insufficiency of the anastomosis will be performed. In case of insufficiency protective ileostomy will be created. 40 patients will be included.

Comparison: Patients with resectable rectal cancer of the middle or lower third will be intraoperatively randomized to either protective ileostomy or no ileostomy at all.

ELIGIBILITY:
Inclusion Criteria:

* radical resectable rectal cancer
* low sphincter-preserving resection of carcinomas of the lower and middle third
* preoperative normal continence
* preoperative normal sphincter function
* complete rings after stapler anastomosis
* impermeability of anastomosis for air
* written informed consent

Exclusion Criteria:

* reduced cooperation or drug abuse
* pregnancy
* psychosis
* age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Morbidity and mortality until day 30 postoperative

SECONDARY OUTCOMES:
Quality of life
Ranking of factors influencing quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Markus W Buchler, Chairman, Principal Investigator — Department of Surgery, University of Heidelberg, Medical School; Peter Kienle, Consultant, Study Chair — Department of Surgery, University of Heidelberg
Locations (1):
- Clinical Study Center Surgery, Department of Surgery, University of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Ulrich AB, Seiler C, Rahbari N, Weitz J, Buchler MW. Diverting stoma after low anterior resection: more arguments in favor. Dis Colon Rectum. 2009 Mar;52(3):412-8. doi: 10.1007/DCR.0b013e318197e1b1. PMID 19333040
- See also: Study Center of the German Surgical Society — http://www.sdgc.de/